CLINICAL TRIAL: NCT04256356
Title: Immunity Modification of Full Term Infants According to the Type of Feeding and Mode of Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heinz Italia SpA (Industry)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FERCT15
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Innate Immunity
Keywords: Newborns; fermented milk; innate immunity
MeSH Terms: interventions — Powders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infants born by CS-fed fermented formula at double dosage (Active Comparator): Infants born by CS-fed formula milk with fermented matrix at dosage of 4,6 g per 100g of powder (group fed with double dosage of fermented matrix compare trial FERCT15)
  Interventions: Dietary Supplement: Feeding infants with formula milk with fermented matrix at dosage of 4.6 g per 100g of powder
- Infants born by CS-fed fermented formula at triple dosage (Active Comparator): Infants born by CS-fed formula milk with fermented matrix at dosage of 6,9 g per 100g of powder (group fed with triple double dosage of fermented matrix compare trial FERCT15)
  Interventions: Dietary Supplement: Feeding infants with formula milk with fermented matrix at dosage of 6.9 g per 100g of powder
- Infants born by CS-fed standard formula (Placebo Comparator): Infants born by CS-fed formula milk without fermented matrix
  Interventions: Other: Feeding infants with standard formula milk
- Infants born by CS-breastfed (Other): Infants born by cesarean section fed with mother milk during were the reference group
  Interventions: Other: Breastfeeding infants

INTERVENTIONS:
Dietary Supplement: Feeding infants with formula milk with fermented matrix at dosage of 4.6 g per 100g of powder — Infants enrolled were fed either with formula milk with fermented matrix at double dosage or with formula milk with fermented matrix at triple dosage or with standard formula during the first 3 months of life. Breastfed infants were the reference group.
  Arms: Infants born by CS-fed fermented formula at double dosage
Dietary Supplement: Feeding infants with formula milk with fermented matrix at dosage of 6.9 g per 100g of powder — Infants enrolled were fed either with formula milk with fermented matrix at double dosage or with formula milk with fermented matrix at triple dosage or with standard formula during the first 3 months of life. Breastfed infants were the reference group.
  Arms: Infants born by CS-fed fermented formula at triple dosage
Other: Feeding infants with standard formula milk — Infants enrolled were fed either with formula milk with fermented matrix at double dosage or with formula milk with fermented matrix at triple dosage or with standard formula during the first 3 months of life. Breastfed infants were the reference group.
  Arms: Infants born by CS-fed standard formula
Other: Breastfeeding infants — reference group
  Arms: Infants born by CS-breastfed

SUMMARY:
This is a single-center, double-blind, randomized controlled trial, with parallel groups and reference group.

The aim of the study was to investigate the immunity of infant born from caesarian section and fed with formula milk containing fermented matrix a double and triple dosage compare the first part of the trial FERCT15 assuming a dose-effect relationship of the fermented matrix with immune response.

DETAILED DESCRIPTION:
The microbiota plays an important role in modulating the development of the immune system, making decisive the interrelation that between nutrition, microbiota and immune cells to modulate long-term health outcomes.

The type of feeding, especially breastfeeding, and the type of delivery are factors that can contribute to the development of the microbiota. Specifically, the exclusive breastfeeding promotes the development of bifidobacteria that promotes protection against potential infections and the development of the immune system.

In recent years it was improved the biological effects of formula milk, that represent the substitutes of breast milk when this is not available or if there are contraindications to breastfeeding. Functional foods derived from fermentation of cow's milk with probiotic strains have been proposed for the prevention of infectious diseases of the child. Recently, in a monocentric double-blind prospective study, the efficacy of fermented cow's milk with Lactobacillus paracasei CBA L74 was evaluated in the prevention of common winter infections in children aged between 12 and 48 months. In this study, children treated with fermented milk had a lower incidence of respiratory and gastrointestinal tract infections compared to the control group. This effect was associated with a significant stimulation of innate immunity (α- and β-defensin, LL-37) and acquired (secretory IgA) and to a modulation of composition and function of the intestinal microbiota characterized by a significant increase in strains producing butyric acid (Firmicutes phyla). The nutritional intervention was very well accepted by the children and no adverse events were observed.

From previous results emerged that in infants born by eutocic delivery fed with fermented formula milk, there is more valid response of innate and acquired immunity compare to controls. In infants born by cesarean section this response is less expressed. It is possible to suppose that this response is linked to a different microbiota.

Primary objectives of this study were:

to investigate the immunity of infant born from caesarian section and fed with formula milk containing fermented matrix a double and triple dosage compare the first part of the trial FERCT15 assuming a dose-effect relationship of the fermented matrix with immune response.

Secondary objective:

Value the tolerance in the two groups of infants fed with the two formulas in the study, with reference to the group of infants fed with breast milk.

Value the modifications of the intestinal microbiota in the 3 groups of infants fed with the 3 formulas in the study, with reference to the group of infants fed with breast milk.

Study design: Single-center, randomized, double-blind, parallel group study with reference group.

Methods:

Evaluation of the anthropometric parameters (weight, length and cranial circumference) Evaluation of body composition by plethysmography Evaluation of the gastrointestinal tolerance of fermented formulated milk by means of data collection and diary delivery to the parents of the participants Evaluation of the safety of fermented formulated milk by recording adverse events Determination of faecal samples of antimicrobial peptides (defensins, catelecidines), IgA, microbiota and metabolome.

Infants will be enrolled at birth (within 7 days of life) upon acquisition of the informed consent of both parents.

At the time of enrollment, infants born by caesarian section who take breast milk due to the absence of breast milk will be randomized to receive up to the third month of age or a standard formula without fermented matrix (control group) or a formula milk containing fermented matrix at dosage of 4.6 g per 100g of powder (group fed with double dosage of fermented matrix compare to FERCT15) or formula milk containing fermented matrix at dosage 6.9 g per 100g of powder (group fed with triple dosage of fermented matrix compare trial FERCT15).

Enrollment will be carried out by promoting and supporting breastfeeding and, in the event of exclusive breastfeeding forecasts for at least the first 3 months of age, newborns will be included in the study as a reference group.

There are 3 medical visits to enrollment (V0), the first (V1) and the third month of life (V2).

During the visits the anthropometric parameters, the body composition, and the gastroenteric tolerance will be evaluated. A stool sample will also be collected at the three points of the life study to determine the anti-microbial peptides (catelecidine, alpha and beta defensin) and the secretory IgA, and perform the analysis of the microbiota and the metabolome.

Statistical analysis:

The sample size was determined considering the secretory IgA values obtained in the FERCT15 trial.

The fecal secretory IgA mean value was 78,3 ±34,37ug/g and of 43,86±30,44 ug/g of feces in the group fed with formula milk with fermented matrix (dosage of 2,3g/100g of powder) and with the standard formula respectively.

Assuming a 15% drop-out rate, 14 newborns per group must be recruited.

Criteria for the evaluation of variables:

The descriptive analyzes will be performed by calculating mean, median and standard deviations for the continuous variables and expressing the distribution of the frequencies for the discrete variables. The main analysis will resort to tests for independent samples, Student or Mann-Whitney tests according to the distribution of the outcome variables. To jointly analyze the trend in time from V0 to V2 of the outcome variables in the two groups, the one that received the fermented formulated milk and the one that received the standard formula, based on the type of delivery (spontaneous or cesarean) will be used regression models for repeated measurements (random effects models or GEE models).

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy infants
* Gestational age from 37 to 41 weeks
* Weight appropriate for gestational age (from 10th to 90th centile according to World Health Organization chart)
* Human milk not available or not possible

Exclusion Criteria:

* Weight small for gestational age (< 10th centile) or large for gestational age (> 90th centile) according to World Health Organization chart
* Congenital abnormalities, chromosomal, hearth, gastrointestinal, respiratory, neurological or metabolic disease.
* Perinatal infections
* Positive familiarity for milk proteins allergies

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Innate immunity at 30 days of life and at 90 days of life. | 0-7 days of life, at 30 days of life and at 90 days of life.
  Fecal dosage of catelecidines, alfa and beta defensins and sIgA

SECONDARY OUTCOMES:
Gastrointestinal tolerance | 0-7 days of life, at 30 days of life and at 90 days of life
  Gastrointestinal tolerance is evaluated by the use of a daily diary computed by the parents to record vomiting/gaseous colics/stool frequency.
Weight | 0-7 days of life, at 30 days of life and at 90 days of life.
  weight (g)
Body composition | Time Frame: 0-7 days of life and at 90 days of life.
  Body composition assessment in term of fat mass and fat free mass by air displacement
Anthropometry | 0-7 days of life, at 30 days of life and at 90 days of life.
  length and head circumference (cm)
Microbiota | 0-7 days of life and at 90 days of life.
  gut microbiota assessment
Metabolomics | 0-7 days of life and at 90 days of life.
  stool metabolomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Mosca, prof, Principal Investigator — NICU. Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not shared with other researchers.

REFERENCES:
- [Background] Zagato E, Mileti E, Massimiliano L, Fasano F, Budelli A, Penna G, Rescigno M. Lactobacillus paracasei CBA L74 metabolic products and fermented milk for infant formula have anti-inflammatory activity on dendritic cells in vitro and protective effects against colitis and an enteric pathogen in vivo. PLoS One. 2014 Feb 10;9(2):e87615. doi: 10.1371/journal.pone.0087615. eCollection 2014. PMID 24520333
- [Background] Thibault H, Aubert-Jacquin C, Goulet O. Effects of long-term consumption of a fermented infant formula (with Bifidobacterium breve c50 and Streptococcus thermophilus 065) on acute diarrhea in healthy infants. J Pediatr Gastroenterol Nutr. 2004 Aug;39(2):147-52. doi: 10.1097/00005176-200408000-00004. PMID 15269618
- [Background] Indrio F, Ladisa G, Mautone A, Montagna O. Effect of a fermented formula on thymus size and stool pH in healthy term infants. Pediatr Res. 2007 Jul;62(1):98-100. doi: 10.1203/pdr.0b013e31806772d3. PMID 17515847
- [Result] Nocerino R, Paparo L, Terrin G, Pezzella V, Amoroso A, Cosenza L, Cecere G, De Marco G, Micillo M, Albano F, Nugnes R, Ferri P, Ciccarelli G, Giaccio G, Spadaro R, Maddalena Y, Berni Canani F, Berni Canani R. Cow's milk and rice fermented with Lactobacillus paracasei CBA L74 prevent infectious diseases in children: A randomized controlled trial. Clin Nutr. 2017 Feb;36(1):118-125. doi: 10.1016/j.clnu.2015.12.004. Epub 2015 Dec 17. PMID 26732025